CLINICAL TRIAL: NCT03509896
Title: Treatment Pattern, Clinical Outcome and Healthcare Resource Utilization Associated With Chinese Newly Diagnosed Patients With Philadelphia Chromosome-Positive (Ph+) Chronic Myeloid Leukemia in Chronic Phase (CML-CP): A Retrospective Observational Study
Brief Title: Study of Chinese Newly Diagnosed Participants With Philadelphia Chromosome-Positive (Ph+) Chronic Myeloid Leukemia in Chronic Phase (CML-CP)
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA180-681
Record Dates: First submitted 2018-04-18; First posted 2018-04-26 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Chronic Myeloid Leukemia; Philadelphia Chromosome; Chronic Myeloid Leukemia in Chronic Phase
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Philadelphia Chromosome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants newly diagnosed with CML-CP
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
Observational medical record review of newly diagnosed CML-CP participants in China

ELIGIBILITY:
Inclusion Criteria:

* Ph+ CML-CP patients who were diagnosed between August 1, 2014 to August 1, 2016
* 18 years or older at time of diagnosis

Exclusion Criteria:

* Participants once enrolled in any interventional clinical trial for CML
* Participants whose records are not available

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multi-center, observational, medical record review of approximately 1000 newly diagnosed CML-CP patients in China
Sampling Method: Probability Sample
Enrollment: 463 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-09-28 (Actual)

PRIMARY OUTCOMES:
Number of participants receiving each first-line treatment option | 2 years
Number of participants with complete cytogenetic response | 2 years
  Complete Cytogenetic Response (CCyR): 0% Ph+ cells in metaphase in bone marrow (BM)
Number of participants with major molecular response (MMR) | 2 years
  Major molecular response (MMR) is defined as 3-log reduction in International Scale of BCR-ABL mRNA
Number of participants of each initial dose schema | 2 years
Starting dose of each first-line agent | 2 years

SECONDARY OUTCOMES:
Distribution of demographic characteristics | 2 years
  Including age, sex, height, weight
Distribution of clinical characteristics | 2 years
  Including health insurance and comorbid conditions

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Tianjin, Tianjin Municipality, China

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm